CLINICAL TRIAL: NCT00250471
Title: A Randomized Trial to Evaluate the Relative Protection Against Post-PCI Microvascular Dysfunction and Post-PCI Ischemia Among Anti-Platelet and Anti-Thrombotic Agents
Brief Title: PROTECT-TIMI 30 Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-046
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2005-11-08 (Estimated); Status verified 2005-11

CONDITIONS: Unstable Angina
Keywords: GP IIb/IIIa inhibitors; eptifibatide; Anti-thrombotic agents
MeSH Terms: conditions — Angina, Unstable | interventions — Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI)

SUMMARY:
The primary purpose of this study was to compare the efficacy and safety of bivalirudin to eptifibatide (with or without unfractionated heparin or enoxaparin)given to subjects at high risk for heart attack and other cardiovascular complications who will undergo surgery to open up blocked arteries in the heart.

DETAILED DESCRIPTION:
Platelet inhibitor drugs

ELIGIBILITY:
Inclusion Criteria:

* Chest paing/discomfort that occurs at rest and lasts at least 10 minutes and have at least one of the following high-risk features:

  * diabetes
  * elevated cardiac proteins in the blood (indicating acute coronary syndrome)
* Be willing and able to give informed consent

Exclusion Criteria:

* uncontrolled hypertension
* cardiac episode (heart attack) within the previous 24 hours before randomization into the trial
* prior heart surgery (PCI) within the previous 2 weeks before randomizing in the trial
* any electorcardogram (ECG) finding that make the Holter monitor for ischemia unable to read

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2003-05; Study Completion 2004-09

PRIMARY OUTCOMES:
Efficacy: Improved Coronary Flow Reserve
Safety: TIMI major hemorrhage within 48 hours after randomizing in the trial or hosptial discharge, which ever occurs first.

SECONDARY OUTCOMES:
Duration of ischemia on continuous EKG monigoring through 24 hours after surgery.
Composite death, heart attack and any occurance of ischemia based on the Holter monitor recording within 48 hours after randomizing into the trial

REFERENCES:
- [Derived] Wilson SR, Sabatine MS, Braunwald E, Sloan S, Murphy SA, Morrow DA. Detection of myocardial injury in patients with unstable angina using a novel nanoparticle cardiac troponin I assay: observations from the PROTECT-TIMI 30 Trial. Am Heart J. 2009 Sep;158(3):386-91. doi: 10.1016/j.ahj.2009.06.011. Epub 2009 Jul 15. PMID 19699861